CLINICAL TRIAL: NCT01093079
Title: Laparoscopic Versus Open Partial Nephrectomy - Surgical and Oncological Outcomes
Acronym: LapVsOpen prtn
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Golan Shay, MD, Rabin Medical Center
Other Study IDs: 5489
Record Dates: First submitted 2010-03-24; First posted 2010-03-25 (Estimated); Last update posted 2010-03-25 (Estimated); Status verified 2009-07

CONDITIONS: Tumor; Nephrectomy; Laparoscopy
Keywords: Renal tumor, RCC, Partial nephrectomy, Laparoscopy
MeSH Terms: conditions — Neoplasms; Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Laparoscopic partial nephrectomy
  Interventions: Procedure: Laparoscopic partial nephrectomy
- Open Partial nephrectomy
  Interventions: Procedure: Open partial nephrectomy

INTERVENTIONS:
Procedure: Laparoscopic partial nephrectomy — Laparoscopic partial nephrectomy
  Groups: Laparoscopic partial nephrectomy
Procedure: Open partial nephrectomy — Open partial nephrectomy
  Groups: Open Partial nephrectomy

SUMMARY:
Partial Nephrectomy is the standard care for small (<4 cm) renal tumors. Despite the expanding use of laparoscopic approach, debate exist regarding the short and long term outcomes compared to the open approach. Our goal is to perform a prospective randomized trial to compare these methods

ELIGIBILITY:
Inclusion Criteria:

* patients referred to partial nephrectomy

Exclusion Criteria:

* Contra-indication for laparocopic surgery
* Complexed , large tumors, single kidney, chronic renal failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred to partial nephrectomy due to renal lesion , suspected to be a tumor
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2009-09

CONTACTS AND LOCATIONS:
Locations (1):
- Rabin medical center, Petah Tikva, Israel